CLINICAL TRIAL: NCT02584881
Title: Safe Opioid Prescription Practice for Patients Discharged From Trauma Services With a Prescription for Opioids
Brief Title: Safe Opioid Prescription Practice for Patients Discharged From Trauma Services
Acronym: SOPP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rhode Island Hospital (Other)
Collaborators: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: U01CE002516-01 (NIH)
Record Dates: First submitted 2014-10-28; First posted 2015-10-23 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2014-10

CONDITIONS: Opioids; Drug Prescription

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): A safe opioid prescription protocol will be implemented with these trauma patients
  Interventions: Other: safe opioid prescription protocol
- Control (No Intervention): Standard care at discharge will be implemented with these trauma patients

INTERVENTIONS:
Other: safe opioid prescription protocol — When indicated a prescription for naloxone will be given to patients discharged with prescription opioids from the trauma services. All patients will receive information on safe opioid use and storage and methods for pain management.
  Arms: Intervention

SUMMARY:
Using a quasi-experimental design the investigators will compare the effect of adopting and implementing a Safe Opioid Prescription Practice (SOPP) protocol within a Level 1 trauma service team compared to a Level 1 trauma service team implementing standard care.

DETAILED DESCRIPTION:
Prescribing opioids to injured patients who are discharged from an inpatient trauma admission is almost ubiquitous; however up to 26% of patients prescribed opioids for chronic pain abuse them leaving them at an increased risk of overdose and overdose fatality. Addressing this problem through an institutional level approach involving both patients and providers, including changes in physician prescription behaviors and directly intervening with the patients to increase knowledge of risks of opioid misuse and overdose, affords us the best opportunity to address this escalating public health concern.

Using a quasi-experimental design the investigators will compare the effect of adopting and implementing a Safe Opioid Prescription Practice (SOPP) protocol within a Level 1 trauma service team compared to a Level 1 trauma service team implementing standard care. Providers at both sites will complete web-based surveys to assess baseline knowledge, attitudes and barriers related to safe prescription practices. The intervention site will complete technical assistance activities to lead to the adoption and implementation of a SOPP protocol. The control site will continue to offer standard care to trauma patients throughout all phases. To measure institutional level changes, chart reviews will be conducted at both sites using a blinded medical review of discharged trauma service patients at baseline, early implementation, implementation and maintenance phases. To measure patient level changes, the investigators will assess patient perception of the discharge experience at both sites during the adoption phase (Cohort 1=100); implementation phase (Cohort 2=100) and maintenance phase (Cohort 3=100) via telephone interview within 7 days post discharge. Three month interviews will also be conducted with Cohort 2 to assess patient opioid usage, pain management strategies and Naloxone usage among Cohort 2. The aims of the proposed research study are to 1) examine and measure the adoption, implementation and maintenance of the SOPP protocol in the intervention site compared to standard care site and 2) to assess patient level outcomes of the SOPP protocol. The secondary aim of this study is to assess the effect the SOPP protocol on provider prescribing practices comparing the average dosage (in morphine milligram equivalents) and duration of dose from the chart review at baseline to the early implementation, implementation and maintenance phases of the study. The findings from this study will allow us to better understand the translation of a safe opioid prescription practice and has the potential to impact best practices for patient discharge within Level 1 trauma centers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Discharged to home from in-patient trauma services with a prescription for opioids
* Responsible for own medication.
* Cognitively capable of giving informed consent, can be contacted by telephone

Exclusion Criteria:

* < 18 years
* Discharged to rehabilitative or nursing home care
* Not discharged with prescribed opioids
* Not responsible for own medication
* No English speaking
* Under arrest at time of in-patient care
* Cannot be contacted by phone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2014-12; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
The frequency of implementation of the SOPP checklist in the intervention site compared to standard care site | Up to 18 months